CLINICAL TRIAL: NCT03245151
Title: A Phase 1/2 Study of Lenvatinib in Combination With Everolimus in Recurrent and Refractory Pediatric Solid Tumors, Including CNS Tumors
Brief Title: Study of Lenvatinib in Combination With Everolimus in Recurrent and Refractory Pediatric Solid Tumors, Including Central Nervous System Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-216
Record Dates: First submitted 2017-08-03; First posted 2017-08-10 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2022-11

CONDITIONS: Recurrent and Refractory Solid Tumors
Keywords: pediatrics; central nervous system tumors; lenvatinib; E7080; everolimus; Ewing sarcoma/peripheral primitive neuroectodermal tumor; rhabdomyosarcoma; high grade glioma; solid tumors
MeSH Terms: conditions — Recurrence; Central Nervous System Neoplasms; Neuroectodermal Tumors, Primitive, Peripheral; Rhabdomyosarcoma; Glioma | interventions — lenvatinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Phase 1; Recurrent or refractory solid tumors (Experimental): During Phase 1 (Treatment Phase: 1 cycle; 28 days of treatment), utilizing a rolling 6 design, participants with recurrent or refractory solid tumors will receive escalating doses of lenvatinib in combination with everolimus for determination of the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D). Participants who complete 1 cycle of treatment will transition to the Extension Phase, in which they will continue to receive the same study treatment in 28-day cycles.
  Interventions: Drug: Lenvatinib; Drug: Everolimus
- Phase 2: Cohort 1, Ewing sarcoma (Experimental): During Phase 2 (four 28-day cycles [up to 16 weeks of treatment]), utilizing Simon's optimal 2-stage design, participants with recurrent or refractory Ewing sarcoma (Cohort 1) will receive the RP2D of lenvatinib in combination with everolimus determined in Phase 1. Participants who discontinue study treatment before completing 4 cycles will transition to the Off-treatment Visit. Participants who complete 4 cycles will transition to the Extension Phase, in which they will continue to receive the same study treatment in 28-day cycles.
  Interventions: Drug: Lenvatinib; Drug: Everolimus
- Phase 2: Cohort 2, Rhabdomyosarcoma (Experimental): During Phase 2 (four 28-day cycles [up to 16 weeks of treatment]), utilizing Simon's optimal 2-stage design, participants with recurrent or refractory rhabdomyosarcoma (Cohort 2) will receive the RP2D of lenvatinib in combination with everolimus determined in Phase 1 (1 cycle; 4 weeks of treatment). Participants who discontinue study treatment before completing 4 cycles will transition to the Off-treatment Visit. Participants who complete 4 cycles will transition to the Extension Phase, in which they will continue to receive the same study treatment in 28-day cycles.
  Interventions: Drug: Lenvatinib; Drug: Everolimus
- Phase 2: Cohort 3, High Grade Glioma (HGG) (Experimental): During Phase 2 (four 28-day cycles [up to 16 weeks of treatment]), utilizing Simon's optimal 2-stage design, participants with recurrent or refractory HGG (Cohort 3) will receive the RP2D of lenvatinib in combination with everolimus determined in Phase 1 (1 cycle; 4 weeks). Participants who discontinue study treatment before completing 4 cycles will transition to the Off-treatment Visit. Participants who complete 4 cycles will transition to the Extension Phase, in which they will continue to receive the same study treatment in 28-day cycles.
  Interventions: Drug: Lenvatinib; Drug: Everolimus

INTERVENTIONS:
Drug: Lenvatinib — oral hard capsules containing 1 mg, 4 mg, or 10 mg lenvatinib, or an extemporaneous suspension
Drug: Everolimus — 2 mg, 3 mg, or 5 mg tablets for oral suspension

SUMMARY:
Phase 1 of this study, utilizing a rolling 6 design, will be conducted to determine a maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D), and to describe the toxicities of lenvatinib administered in combination with everolimus once daily to pediatric participants with recurrent/refractory solid tumors. Phase 2, utilizing Simon's optimal 2-stage design, will be conducted to estimate the antitumor activity of lenvatinib in combination with everolimus in pediatric participants with selected recurrent/refractory solid tumors including Ewing sarcoma, rhabdomyosarcoma, and high grade glioma (HGG) using objective response rate (ORR) at Week 16 as the outcome measure.

ELIGIBILITY:
Inclusion Criteria

* ≥2 years and <18 years of age for enrolment in Phase 1 or ≥2 years and ≤21 years of age for enrolment in Phase 2.
* Recurrent or refractory solid tumors

  * Phase 1: All solid tumors (measurable or evaluable disease), including primary central nervous system (CNS) tumors; exclusion of hepatoblastoma and lymphomas. Participants with diffuse intrinsic pontine glioma, optic pathway glioma, or pineal tumors with elevated tumor markers (alpha-fetoprotein [AFP] and beta-human chorionic gonadotropin [ß-hCG][or human chorionic gonadotropin [hCG])do not require histological or cytological confirmation of diagnosis
  * Phase 2: Ewing sarcoma, Rhabdomyosarcoma, High Grade Glioma (HGG) (all must have measurable disease); exclusion of Diffuse Intrinsic Pontine Glioma
* Histologically or cytologically confirmed diagnosis
* Measurable disease that meets the following criteria (Phase 2):

  1. RECIST 1.1 (for all tumor types except HGG): At least 1 lesion of ≥1.0 cm in the longest diameter for a non lymph node or ≥1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computed tomography /magnetic resonance imaging (CT/MRI)
  2. Response Assessment in Neuro-Oncology (RANO) for high grade glioma (HGG): At least one lesion must be measurable as defined as a bi dimensionally contrast enhancing lesion with clearly defined margins by CT or MRI scan, with a minimal diameter of 1 cm, and visible on 2 axial slices which are preferably at most 5 mm apart with 0 mm skip

Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion

* Karnofsky performance score ≥50 for participants>16 year of age and Lansky play score ≥50 for participants ≤16 years of age. Neurologic deficits in participants with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Prior Therapy

  * Participants must have fully recovered from the acute toxic effects of all prior anti-cancer therapy
  * Cytotoxic chemotherapy or other chemotherapy known to be myelosuppressive: ≥21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (eg, not associated with reduced platelet or absolute neutrophil counts): ≥7 days after the last dose of agent
  * Monoclonal antibodies: ≥21 days or 3 half-lives (whichever is shorter) of the antibody must have elapsed after the last dose of a monoclonal antibody (including checkpoint inhibitors). Toxicity related to prior antibody therapy must be recovered to Grade ≤1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, ≥14 days must have elapsed since last dose of corticosteroid. Participants receiving corticosteroids, who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment, are not eligible
  * Hematopoietic growth factors: ≥14 days after the last dose of a long-acting growth factor or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Interleukins, interferons, and cytokines (other than hematopoietic growth factors): ≥21 days after the completion of interleukins, interferons or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without total body irradiation): Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor leukocytes infusion or boost infusion: ≥84 days after infusion and no evidence of graft versus host disease; Autologous stem cell infusion including boost infusion: ≥42 days
  * Cellular Therapy: ≥42 days after the completion of any type of cellular therapy (eg, modified T cells, natural killer cells, dendritic cells, etc)
  * Radiotherapy (XRT)/External Beam Irradiation including Protons: ≥14 days after local XRT; ≥150 days after total body irradiation, craniospinal XRT or if radiation to ≥50% of the pelvis; ≥42 days if other substantial bone marrow radiation.
  * Radiopharmaceutical therapy: ≥42 days after systemically administered therapy.
  * Vascular endothelial growth factor (VEGF)/VEGF receptor (VEGFR)-targeted or mammalian target of rapamycin (mTOR)-targeted therapies: Must not have received prior exposure to lenvatinib; May have previously progressed on an mTOR inhibitor; No more than 2 prior VEGF/VEGFR-targeted therapies (For Phase 2 only); Must not have received prior VEGF/VEGFR-targeted therapy in combination with an mTOR inhibitor (For Phase 2 only)
* Adequate bone marrow function for participants with solid tumors without known bone marrow involvement
* Adequate bone marrow function for participants with known bone marrow metastatic disease
* Adequate renal function
* Adequate liver function
* Adequate cardiac function
* Adequate neurologic function
* Adequate blood pressure (BP) control with or without antihypertensive medications
* Adequate coagulation
* Adequate pancreatic function
* Adequate metabolic function
* Adequate glycemic control
* Participants must have a minimum body surface area (BSA) of 0.6 m^2 at study entry.

Exclusion Criteria

* Participants who have had or are planning to have the following invasive procedures

  * Major surgical procedure, laparoscopic procedure, open biopsy or significant traumatic injury within 28 days prior to enrolment
  * Central line placement or subcutaneous port placement is not considered major surgery. External central lines must be placed at least 3 days prior to enrollment and subcutaneous ports must be placed at least 7 days prior to enrollment
  * Fine needle aspirate within 7 days prior to enrolment
  * Surgical or other wounds must be adequately healed prior to enrolment
  * For purposes of this study, bone marrow aspirate and biopsy are not considered surgical procedures and therefore are permitted within 14 days prior to start of protocol therapy
* Participants who have non-healing wound, unhealed or incompletely healed fracture, or a compound (open) bone fracture at the time of enrolment
* Participants having an active infection requiring systemic therapy.
* Participants with a known history of active hepatitis B (defined as hepatitis B surface antigen reactive or hepatitis B virus- deoxyribonucleic [DNA] detected) or known active hepatitis C virus (HCV, defined as HCV- Ribonucleic acid [RNA] detected). Note: No testing for hepatitis B and hepatitis C is required unless mandated by the local health authority.
* Known to be human immunodeficiency virus (HIV) positive. Note: HIV testing is required at screening only when mandated by the local health authority
* Clinical evidence of nephrotic syndrome prior to enrolment
* Gastrointestinal bleeding or active hemoptysis (bright red blood of at least half teaspoon) within 21 days prior to enrolment
* Thrombotic/ thromboembolic event requiring systemic anticoagulation within 90 days prior to enrollment
* Evidence of new intracranial hemorrhage of more than punctate size on MRI assessment obtained within 28 days prior to study enrollment for Participants with HGG
* Diagnosis of lymphoma
* Radiographic evidence of major blood vessel invasion/infiltration.
* Evidence of untreated CNS metastases (exception: participants with primary CNS tumors and leptomeningeal disease)
* Participants who are currently receiving enzyme-inducing anticonvulsants
* Participants chronically receiving strong cytochrome P450 3A4 (CYP3A4)/P-glycoprotein (P-gp) inhibitors or inducers within 7 days prior to study enrollment
* Females who are breastfeeding or pregnant. For females of childbearing potential, a negative screening pregnancy test must be obtained within 72 hours before the first dose of study drug
* Males who have not had a successful vasectomy (confirmed azoospermia) or if they and their female partners do not meet the criteria above (that is, not of childbearing potential or practicing highly effective contraception throughout the study period and for 7 days after lenvatinib discontinuation or 4 weeks after discontinuation of everolimus). No sperm donation is allowed during the study period and for 7 days after lenvatinib discontinuation or 4 weeks after discontinuation of everolimus.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (47):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital, Long Beach, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Kaiser Permenente, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center at Mission Bay - Pediatric Oncology, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours/ Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Kapi'olani Medical Center, Honolulu, Hawaii
  - St Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children - Indiana University, Indianapolis, Indiana
  - University of Louisville and Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Alliance for Childhood Diseases, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers cancer Institute of NJ, New Brunswick, New Jersey
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - The Children's Hospital of San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Dela Cruz FS, Fox E, DuBois SG, Friedman GK, Croop JM, Kim A, Morgenstern DA, Balis FM, Macy ME, Pressey JG, Watt T, Krystal JI, Vo KT, Mody R, Laetsch TW, Weigel BJ, O'Hara K, He CS, Aluri J, Okpara CE, Glade Bender JL. A Phase 1/2 Study of Lenvatinib in Combination With Everolimus in Recurrent and Refractory Pediatric and Young Adult Solid Tumors. Pediatr Blood Cancer. 2025 Jul;72(7):e31692. doi: 10.1002/pbc.31692. Epub 2025 May 1. PMID 40313040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 24 investigative sites in the United States and Canada from 16 November 2017 to 30 September 2022.
Pre-assignment Details: A total of 86 participants were screened, out of which 64 were enrolled and 9 participants completed the study.
Groups:
- Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2: Participants with recurrent or refractory solid tumors received lenvatinib 8 milligram per square meter (mg/m^2), capsules, orally, once daily in combination with everolimus 3 mg/m^2, tablets, orally, once daily in cycle 1 (each cycle was 28 days) until the occurrence of disease progression (PD), clinical benefit, development of unacceptable toxicity leading to withdrawal from the study, study discontinuation or for a maximum of 18 cycles (each cycle was 28 days) whichever occurred first.
- Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2: Participants with recurrent or refractory solid tumors received lenvatinib 11 mg/m^2, capsules, orally, once daily in combination with everolimus 3 mg/m^2, tablets, orally, once daily in cycle 1 (each cycle was 28 days) until the occurrence of PD, clinical benefit, development of unacceptable toxicity leading to withdrawal from the study, study discontinuation or for a maximum of 18 cycles (each cycle was 28 days) whichever occurred first.
- Phase 2: Cohort 1, Ewing Sarcoma: Participants with recurrent or refractory ewing sarcoma received lenvatinib 11 mg/m^2, capsules, orally, once daily in combination with everolimus 3 mg/m^2, tablets, orally, once daily for up to 7 cycles (each cycle was 28 days) unless participant discontinued early from the study.
- Phase 2: Cohort 2, Rhabdomyosarcoma: Participants with recurrent or refractory rhabdomyosarcoma received lenvatinib 11 mg/m^2, capsules, orally, once daily in combination with everolimus 3 mg/m^2, tablets, orally, once daily for up to 7 cycles (each cycle was 28 days) unless participant discontinued early from the study.
- Phase 2: Cohort 3, HGG: Participants with recurrent or refractory high grade glioma (HGG) received lenvatinib 11 mg/m^2, capsules, orally, once daily in combination with everolimus 3 mg/m^2, tablets, orally, once daily for up to 7 cycles (each cycle was 28 days) unless participant discontinued early from the study.
Period: Overall Study
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2 | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
Started | 5 | 18 | 10 | 20 | 11
Completed | 0 | 3 | 1 | 2 | 3
Not Completed | 5 | 15 | 9 | 18 | 8
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 1
Not completed — Death | 3 | 14 | 9 | 16 | 7
Not completed — Sponsor's decision | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants who received at least 1 dose of study drug (lenvatinib or everolimus).
Groups:
- Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2: Participants with recurrent or refractory solid tumors received lenvatinib 8 mg/m^2, capsules, orally, once daily in combination with everolimus 3 mg/m^2, tablets, orally, once daily in cycle 1 (each cycle was 28 days) until the occurrence of PD, clinical benefit, development of unacceptable toxicity leading to withdrawal from the study, study discontinuation or for a maximum of 18 cycles (each cycle was 28 days) whichever occurred first.
- Phase 2: Cohort 3, HGG: Participants with recurrent or refractory HGG received lenvatinib 11 mg/m^2, capsules, orally, once daily in combination with everolimus 3 mg/m^2, tablets, orally, once daily for up to 7 cycles (each cycle was 28 days) unless participant discontinued early from the study.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2 | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG | Total
Number analyzed (Participants) | 5 | 18 | 10 | 20 | 11 | 64
Age, Customized [Count of Participants; unit: Participants]
  2-11 years | 0 | 16 | 3 | 9 | 3 | 31
  12-17 years | 4 | 1 | 3 | 6 | 7 | 21
  18-64 years | 1 | 1 | 4 | 5 | 1 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 3 | 8 | 8 | 31
  Male | 3 | 8 | 7 | 12 | 3 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 2 | 2 | 0 | 12
  Not Hispanic or Latino | 4 | 11 | 8 | 18 | 11 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 3 | 6
  White | 3 | 11 | 9 | 16 | 6 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 0 | 3 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Lenvatinib in Combination With Everolimus
Description: MTD was defined as the highest dose level at which no more than 1/6 participants experienced a dose limiting toxicity (DLTs), with the next higher dose having at least 0 of 3 or 1 of 6 participants experiencing DLTs. DLT was graded according to common terminology criteria for adverse events (CTCAE) version 4.03.
Time Frame: Cycle 1 (Each cycle was of 28 days)
Population: SAS included all participants who received at least one dose of study drug (Lenvatinib or Everolimus).
Measure: Number; unit: milligram per square meter (mg/m^2)
Groups:
- Phase 1: Lenvatinib + Everolimus (All Participants): Participants with recurrent or refractory solid tumors received lenvatinib 8 or 11 mg/m^2, capsules, orally, once daily in combination with everolimus 3 mg/m^2, tablets, orally, once daily in cycle 1 (each cycle was 28 days) until the occurrence of PD, clinical benefit, development of unacceptable toxicity leading to withdrawal from the study, study discontinuation or for a maximum of 18 cycles (each cycle was 28 days) whichever occurred first.
Arm/Group | Phase 1: Lenvatinib + Everolimus (All Participants)
Number analyzed (Participants) | 23
milligram per square meter (mg/m^2) | 11

2. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D) of Lenvatinib in Combination With Everolimus
Description: The RP2D of lenvatinib in combination with everolimus was determined by Dose Escalation Committee (DEC) based on safety (including DLTs), pharmacokinetic and clinical data. DLT was graded according to CTCAE v4.03.
Time Frame: Cycle 1 (Each cycle was of 28 days)
Population: SAS included all participants who received at least one dose of study drug (Lenvatinib or Everolimus).
Measure: Number; unit: mg/m^2
Arm/Group | Phase 1: Lenvatinib + Everolimus (All Participants)
Number analyzed (Participants) | 23
mg/m^2 | 11

3. Primary Outcome: Phase 1: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an adverse event that emerged during treatment, having been absent at pretreatment or reemerged during treatment, having been present at pretreatment but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the adverse event is continuous. An adverse event was defined as any untoward medical occurrence in a participant administered an investigational product.
Time Frame: From date of first dose up to 28 days after the last dose of study treatment (Up to 17.5 months)
Population: SAS included all participants who received at least one dose of study drug (Lenvatinib or Everolimus).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 5 | 18
Participants | 5 | 18

4. Primary Outcome: Phase 1: Number of Participants With Any Treatment-emergent Serious Adverse Event (TESAE)
Description: A TESAE was any untoward medical occurrence that at any dose: resulted in death; life threatening condition; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or was medically important due to other reasons than the above mentioned criteria. An adverse event was defined as any untoward medical occurrence in a participant administered an investigational product.
Time Frame: From date of first dose up to 28 days after the last dose of study treatment (Up to 17.5 months)
Population: SAS included all participants who received at least one dose of study drug (Lenvatinib or Everolimus).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 5 | 18
Participants | 2 | 12

5. Primary Outcome: Phase 2: Objective Response Rate (ORR) at Week 16
Description: ORR at Week 16 was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) at Week 16 based on investigator assessment according to response evaluation criteria in solid tumors (RECIST) version 1.1 for non-HGG cohorts and response assessment in neuro-oncology (RANO) for HGG cohort. CR was defined as disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis less than (<) 10 millimeter (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameter (SOD) of target lesions, taking as reference the baseline sum diameters.
Time Frame: Week 16
Population: Evaluable analysis set included all evaluable participants who have measurable disease present at baseline, and at least one postbaseline efficacy assessment, unless they have discontinued prior to the first efficacy assessment due to progressive disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
Number analyzed (Participants) | 10 | 20 | 10
percentage of participants | 0.0 (0.0) [0.0 to 30.8] | 10.0 (1.2) [1.2 to 31.7] | 0 (0.0) [0.0 to 30.8]

6. Secondary Outcome: Phase 1: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with BOR of CR or PR based on investigator assessment according to RECIST version 1.1 for non-HGG cohorts and RANO for HGG cohort. CR was defined as disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of the first dose of study drug to the date of first documentation of disease progression or death, whichever occurred first (up to 16.5 months)
Population: SAS included all participants who received at least 1 dose of study drug (lenvatinib or everolimus). Here, 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 3 | 15
percentage of participants | 0.0 (0.0) [0.0 to 70.8] | 0.0 (0.0) [0.0 to 21.8]

7. Secondary Outcome: Phase 2: Objective Response Rate (ORR)
Description: as for outcome 6
Time Frame: From the date of the first dose of study drug to the date of first documentation of disease progression or death, which ever occurred first (up to 6.5 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
Number analyzed (Participants) | 10 | 20 | 10
percentage of participants | 0.0 (0.0) [0.0 to 30.8] | 10.0 (1.2) [1.2 to 31.7] | 0.0 (0.0) [0.0 to 30.8]

8. Secondary Outcome: Phase 1: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with a confirmed CR, PR, or stable disease (SD) (SD duration >=7 weeks since the first dose of study treatment) divided by number of participants in analysis set. DCR was assessed by an investigator based on RECIST v1.1 for non-HGG participants or RANO for HGG participants. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From first dose of study drug until PD or death, whichever occurred first (up to 16.5 months)
Population: SAS included all participants who received at least 1 dose of study drug (lenvatinib or everolimus).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 5 | 18
percentage of participants | 20.0 (0.5) [0.5 to 71.6] | 50.0 (26.0) [26.0 to 74.0]

9. Secondary Outcome: Phase 2: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with confirmed CR, PR, or SD (SD duration greater than or equal to [>=] 7 weeks since first dose of study treatment) divided by number of participants in analysis set. DCR was assessed by investigator based on RECIST v1.1 for non-HGG cohorts or RANO for HGG cohort. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From first dose of study drug until PD or death, whichever occurred first (up to 6.5 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
Number analyzed (Participants) | 10 | 20 | 10
percentage of participants | 40.0 (12.2) [12.2 to 73.8] | 40.0 (19.1) [19.1 to 63.9] | 30.0 (6.7) [6.7 to 65.2]

10. Secondary Outcome: Phase 1: Clinical Benefit Rate (CBR)
Description: CBR was defined as percentage of participants who had BOR of CR, PR, or durable SD (SD duration >=23 weeks since the first dose of study treatment) divided by number of participants in analysis set. CBR was assessed by an investigator based on RECIST v1.1 for non-HGG participants or RANO for HGG participants. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From first dose of study drug until PD or death, whichever occurred first (up to 16.5 months)
Population: SAS included all participants who received at least 1 dose of study drug (lenvatinib or everolimus).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 5 | 18
percentage of participants | 20.0 (0.5) [0.5 to 71.6] | 22.2 (6.4) [6.4 to 47.6]

11. Secondary Outcome: Phase 2: Clinical Benefit Rate (CBR)
Description: CBR was defined as percentage of participants who had BOR of CR, PR, or durable SD (SD duration >=23 weeks since the first dose of study treatment) divided by number of participants in analysis set. CBR was assessed by an investigator based on RECIST v1.1 for non-HGG cohorts or RANO for HGG cohort. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From first dose of study drug until PD or death, whichever occurred first (up to 6.5 months)
Population: Evaluable analysis set included all evaluable participants who have measurable disease present at baseline, and at least one postbaseline efficacy assessment, unless they have discontinued prior to the first efficacy assessment due to PD.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
Number analyzed (Participants) | 10 | 20 | 10
percentage of participants | 20.0 (2.5) [2.5 to 55.6] | 10.0 (1.2) [1.2 to 31.7] | 0.0 (0.0) [0.0 to 30.8]

12. Secondary Outcome: Phase 1: Duration of Response (DOR)
Description: DOR was defined as the time (in months) from the date of first observation of confirmed response (PR or CR) to the date of the first observation of progression based on the investigator's assessment utilizing RECIST 1.1 for non-HGG cohorts and RANO for HGG cohorts, or date of death, whatever the cause. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From date of the first observation of CR or PR until the date of first observation of progression or date of death (up to 16.5 months)
Population: SAS included all participants who received at least 1 dose of study drug (lenvatinib or everolimus). Here, 'overall number of participants analyzed' signifies participants who had CR or PR (0 participants hence, none were analyzed for this outcome measure).
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was defined as the time (in months) from the date of first observation of confirmed response (PR or CR) to the date of the first observation of progression based on the investigator's assessment utilizing RECIST 1.1 for non-HGG cohorts and RANO for HGG cohort, or date of death, whatever the cause. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From date of the first observation of CR or PR until the date of first observation of progression or date of death (up to 6.5 months)
Population: Evaluable analysis set included all evaluable participants who have measurable disease present at baseline, and at least one postbaseline efficacy assessment, unless they have discontinued prior to first efficacy assessment due to progressive disease. Here, 'overall number of participants analyzed' signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
Number analyzed (Participants) | 0 | 2 | 0
months |  | 2.4 [2.1 to NA] — Upper limit of 95% Confidence Interval could not be estimated as insufficient number of participants were available for analysis. |

14. Secondary Outcome: Phase 1: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration of Lenvatinib (AUC[0-t Hours])
Description: AUC0-t of lenvatinib was quantified using validated liquid chromatography tandem mass spectrometry (LC-MS/MS) methods.
Time Frame: Cycle 1 Days 1 and 15: 0-8 hours post-dose (Cycle length=28 days)
Population: Pharmacokinetic analysis set included participants who had at least one measurable postdose plasma concentration with an adequately documented drug administration history. Here, 'number analyzed' signifies participants who were evaluable for given timepoints of this outcome measure. Pharmacokinetic data was planned to be analyzed for Phase 1 only.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 5 | 18
nanogram*hour per milliliter (ng*hr/mL)
  Cycle 1 Day 1 | 2338.0 (1633.41) | 3281.1 (1064.72)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 17
  Cycle 1 Day 15 | 1328.0 (520.69) | 2139.8 (1156.48)

15. Secondary Outcome: Phase 1: Maximum Plasma Concentration of Lenvatinib (Cmax)
Description: Cmax of lenvatinib was quantified using validated liquid LC-MS/MS methods.
Time Frame: Cycle 1 Days 1 and 15: 0-8 hours post-dose (Cycle length=28 days)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 5 | 18
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 240.20 (130.892) | 404.13 (121.473)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 17
  Cycle 1 Day 15 | 314.20 (149.527) | 447.62 (272.790)

16. Secondary Outcome: Phase 1: Time to Reach Maximum Plasma Concentration (Cmax) of Lenvatinib (Tmax)
Description: Tmax of lenvatinib was quantified using validated liquid LC-MS/MS methods.
Time Frame: Cycle 1 Days 1 and 15: 0-8 hours post-dose (Cycle length=28 days)
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 5 | 18
hours
  Cycle 1 Day 1 | 3.000 [2.000 to 4.000] | 2.890 [1.000 to 7.78]
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 17
  Cycle 1 Day 15 | 3.950 [2.000 to 8.05] | 2.950 [0 to 8.02]

17. Secondary Outcome: Phase 1: Trough Concentrations (Ctrough) of Everolimus When Administered in Combination With Lenvatinib
Description: Trough concentrations of everolimus was quantified using validated liquid LC-MS/MS methods.
Time Frame: Cycle 1 Days 1, 2, 15 and 22: Pre-dose (Cycle length=28 days)
Population: Pharmacokinetic analysis set included participants who had at least one measurable postdose plasma concentration with an adequately documented drug administration history. Here, 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and 'number analyzed' signifies participants who were evaluable for given timepoints of this outcome measure. Pharmacokinetic data was planned to be analyzed for Phase 1 only.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2
Number analyzed (Participants) | 5 | 17
ng/mL
  Cycle 1 Day 1: Pre-dose | 0.0 (0.0) | 0.0 (0.00)
  Cycle 1 Day 2: Pre-dose | 2.1 (1.34) | 2.2 (1.13)
  Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 5 | 15
  Cycle 1 Day 15: Pre-dose | 3.2 (2.42) | 5.1 (2.98)
  Cycle 1 Day 22: Pre-dose: number analyzed (Participants) | 5 | 15
  Cycle 1 Day 22: Pre-dose | 2.8 (1.96) | 4.2 (2.73)

18. Secondary Outcome: Phase 2: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: as for outcome 3
Time Frame: From date of first dose up to 28 days after the last dose of study treatment (up to 7.5 months)
Population: SAS included all participants who received at least one dose of study drug (Lenvatinib or Everolimus).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
Number analyzed (Participants) | 10 | 20 | 11
Participants | 10 | 19 | 11

19. Secondary Outcome: Phase 2: Number of Participants With Any Treatment-emergent Serious Adverse Event (TESAE)
Description: as for outcome 4
Time Frame: From date of first dose up to 28 days after the last dose of study treatment (up to 7.5 months)
Population: SAS included all participants who received at least one dose of study drug (Lenvatinib or Everolimus).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
Number analyzed (Participants) | 10 | 20 | 11
Participants | 6 | 8 | 8

ADVERSE EVENTS:
Time Frame: From date of first dose up to 28 days after the last dose of study treatment (Phase 1: Up to 17.5 months; Phase 2: Up to 7.5 months)
Description: SAS included all participants who received at least 1 dose of study drug (lenvatinib or everolimus).
Arm/Group | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2 | Phase 2: Cohort 1, Ewing Sarcoma | Phase 2: Cohort 2, Rhabdomyosarcoma | Phase 2: Cohort 3, HGG
All-Cause Mortality (participants affected / at risk) | 4/5 | 14/18 | 9/10 | 17/20 | 8/11
Serious Adverse Events (participants affected / at risk) | 2/5 | 12/18 | 6/10 | 8/20 | 8/11
Other Adverse Events (participants affected / at risk) | 5/5 | 18/18 | 10/10 | 19/20 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 (N=5) | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2 (N=18) | Phase 2: Cohort 1, Ewing Sarcoma (N=10) | Phase 2: Cohort 2, Rhabdomyosarcoma (N=20) | Phase 2: Cohort 3, HGG (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infections (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral cavity fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Lenvatinib 8 mg/m^2 + Everolimus 3 mg/m^2 (N=5) | Phase 1: Lenvatinib 11 mg/m^2 + Everolimus 3 mg/m^2 (N=18) | Phase 2: Cohort 1, Ewing Sarcoma (N=10) | Phase 2: Cohort 2, Rhabdomyosarcoma (N=20) | Phase 2: Cohort 3, HGG (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 (6) | 6 (16) | 5 (17) | 7 (10) | 1 (5)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (6) | 4 (5) | 1 (2) | 3 (5) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3) | 10 (13) | 2 (3) | 8 (14) | 6 (7)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 9 (16) | 1 (1) | 7 (10) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 3 (4) | 4 (5) | 6 (8) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (10) | 10 (23) | 5 (10) | 8 (11) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (9) | 5 (8) | 3 (4) | 9 (14) | 4 (5)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (10) | 5 (8) | 2 (2) | 9 (21) | 2 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (10) | 11 (20) | 3 (7) | 7 (11) | 7 (10)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 6 (9) | 6 (7) | 11 (16) | 3 (5)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 5 (7) | 4 (8) | 3 (4) | 0 (0)
Pain (General disorders) | 3 (7) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Malaise (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (7) | 1 (1) | 5 (8) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gait disturbances (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infections (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (10) | 3 (7) | 7 (7) | 3 (4)
Amylase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 5 (13) | 4 (6) | 8 (13) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (3)
Blood cholesterol increased (Investigations) | 1 (1) | 6 (23) | 2 (2) | 11 (14) | 4 (12)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (4) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 3 (9) | 3 (5)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (14) | 6 (13) | 8 (27) | 11 (32) | 2 (10)
Neutrophil count decreased (Investigations) | 3 (6) | 4 (12) | 3 (7) | 7 (14) | 2 (9)
Platelet count decreased (Investigations) | 2 (6) | 7 (22) | 5 (9) | 10 (21) | 3 (4)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (3) | 6 (12) | 1 (2) | 6 (10) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3)
White blood cell count decreased (Investigations) | 2 (7) | 6 (16) | 6 (17) | 8 (24) | 2 (8)
Decreased appetite (Metabolism and nutrition disorders) | 4 (7) | 4 (5) | 2 (3) | 6 (9) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (5) | 1 (2) | 4 (5) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 2 (2) | 4 (6) | 3 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (4) | 3 (6) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (3) | 11 (51) | 5 (18) | 12 (26) | 6 (22)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (9) | 5 (13) | 4 (14) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 5 (7) | 4 (6) | 0 (0)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (6) | 2 (2) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 6 (7) | 7 (15) | 2 (3) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (6) | 8 (14) | 6 (10) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (3) | 3 (5) | 6 (11) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 4 (6) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (5) | 1 (5) | 4 (6) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (9) | 2 (2) | 5 (7) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrous cortical defect (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) | 1 (3) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (14) | 8 (10) | 1 (1) | 5 (5) | 5 (7)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 2 (3) | 2 (2) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (4) | 8 (37) | 8 (15) | 10 (23) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 4 (5) | 6 (6) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal tubular dysfunction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7) | 1 (1) | 4 (5) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 2 (2) | 4 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (9) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 1 (1) | 5 (5) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (3) | 7 (12) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (5) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 1 (1) | 2 (4) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6) | 0 (0) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (5) | 2 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6) | 0 (0) | 3 (4) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (14) | 13 (19) | 3 (4) | 10 (18) | 4 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 2 (4) | 1 (1) | 2 (2) | 1 (1)
Erythemas (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT03245151/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT03245151/SAP_001.pdf